CLINICAL TRIAL: NCT06482619
Title: Effects of Creatine Supplementation in Combination With a Rehabilitation Program Physical in Athletes With Patellar Tendinopathy
Brief Title: Effects of Creatine and Rehabilitation Programin Athletes With Patellar Tendinopathy
Acronym: CREATINE_TEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Pontificia Comillas (Other)
Collaborators: Universidad de Córdoba (Other); University of Bologna (Other); Technical University of Madrid (Other); Lavras University (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UPComillas
Record Dates: First submitted 2024-06-25; First posted 2024-07-01 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Creatine; Patellar Tendinopathy
Keywords: Ergogenic aid; Dietary; Injury; Nutrition; Sport Nutrition
MeSH Terms: conditions — Wounds and Injuries | interventions — Creatine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A researcher who did not have any contact with the participants and the physiotherapist who performed the physical rehabilitation intervention and the assessments randomly divided the participants to the creatine or placebo groups in a computerized random list with a 1:1 allocation using the software Research Randomizer (www.randomizer.org).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Creatine supplementation (Experimental): Creatine monohydrate (Creapure®, Crown Sport Nutrition, Arnedo, Spain) ingested 3 capsules daily (3 g/day)
  Interventions: Dietary Supplement: Creatine supplementation
- Placebo supplementation (Placebo Comparator): Sucrose ingested 3 capsules daily (3 g/day)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Creatine supplementation — The supplements were provided in capsules of 1 g of red color not transparent Guinama S.L.U, 0044634, La Pobla de Valbona, Spain) which were prepared with a Capsunorm 2000 semi-automatic manual capsule filling machine (Miranda del Ebro, Spain). Capsules contained creatine monohidrate (Creapure, Crown Sport Nutrition, Arnedo, Spain)
  Arms: Creatine supplementation
Dietary Supplement: Placebo — The supplements were provided in capsules of 1 g of red color not transparent Guinama S.L.U, 0044634, La Pobla de Valbona, Spain) which were prepared with a Capsunorm 2000 semi-automatic manual capsule filling machine (Miranda del Ebro, Spain). Capsules contained placebo (i.e., sucrose)
  Arms: Placebo supplementation

SUMMARY:
The aim of this study are to analyze the effect of creatine ingestion in pain, histological properties of the tendon, body composition, strength and vertical jump performance in athletes with patellar tendinopathy that follow a physical rehabilitation program that include eccentric exercise combined with stretching and extracorporeal shock wave therapy.

DETAILED DESCRIPTION:
Nutrition could play an important role in the rehabilitation from sport injuries. This afirmation is based on studies that analyze the impact of different dietary supplements along immobilization periods, stablishing that creatine, leucine and omega-3 fatty acid supplementation could ameliorate muscle loss, while creatine could potentiate the hypertrophy along the rehabilitation process. For this reason, the aim of this study are to analyze the effect of creatine ingestion in pain, histological properties of the tendon, body composition, strength and vertical jump performance in athletes with patellar tendinopathy that follow a physical rehabilitation program that include eccentric exercise combined with stretching and extracorporeal shock wave therapy.

ELIGIBILITY:
Inclusion Criteria:

* Athletes diagnosed with patellar tendinopathy by sport medicine doctor.
* Age (>18 years and <49 years).
* To be federated in a sport modality that involves high repetitive impact in the knee; iii) to train more than 3 sessions weekly.
* Not having undergone knee surgery.
* Not having undergone any infiltration of analgesics or platelet-rich plasma during the last year.
* Not intake any sport performance supplement in the previous year;
* Smoker person.

Exclusion Criteria:

* Not being diagnosed with patellar tendinopathy by a doctor
* Age (<18 years and > 50 years).
* Involved in a sport modality without high repetitive impacts during sports activity.

Ages: 18 Years to 49 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Pain evaluation | 8-weeks
  For assessing pain, the Victorian Institute for Sports Assessment - Patella (VISA - P), the most widely used patient-reported outcome measure (including symptom severity), was administered . The VISA - P will be scored with a maximum of 100 points and the higher scores indicate better function, and it shows sensible to identify improvements in therapeutic interventions among patients with tendinopathies.
Tendon thickness. | 8-weeks
  Thickness Tendon of the injuried knee/s was analyzed with ultrasound (GE VENUE 40, Portable Ultrasound, CA, USA), and a linear translator. Participants were positioned supine with a 30º knee flexion (using a roller under the knees), reducing the "locking" of the patella in the femur as in full extension. Ultrasound gel was applied and evaluated by placing the probe longitudinally; in pathological tendons it is the only way to determine the distance of the measurement point from the insertion of the tendon. Thus, subsequent measurements were always made from the same point.

SECONDARY OUTCOMES:
Neuromuscular function | 8-weeks
  Participants performed a neuromuscular test battery consisted in measuring vertical jump capacity (i.e., countermovement jump) and knee extension muscle strength muscular strength in a knee extension machine (Selection Leg Extension, Technogym, Cesena, Italy) with a 5 maximum number of repetitions (5-RM)

CONTACTS AND LOCATIONS:
Overall Officials: Angela Sánchez-Gómez, PhD, Principal Investigator — Universidad de Córdoba
Locations (1):
- Universidad Pontificia Comillas, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No